CLINICAL TRIAL: NCT05040659
Title: Longitudinal At Home Smell Testing to Detect Infection by SARS-CoV-2
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Mark W Albers, Frank Wilkens and Family Endowed Scholar/ Asst. Prof. Neurology, Massachusetts General Hospital
Other Study IDs: 2021P001988; U01DC019579 (NIH)
Record Dates: First submitted 2021-08-18; First posted 2021-09-10 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Anosmia; Asymptomatic COVID-19; COVID-19 Respiratory Infection; Influenza; Healthy; PASC Post Acute Sequelae of COVID 19
MeSH Terms: conditions — Anosmia; Influenza, Human; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Anosmic patients: Anosmic patients will be recruited from Dr. Albers Smell Clinic at MGH and through past participation in research with known anosmia and permission to recontact. All consent and testing will occur on a phone/tablet app in the participant's home.
  Interventions: Device: AROMHA Longitudinal Smell Test
- Asymptomatic participants / Healthy participants: Asymptomatic participants recruited in a hospital setting (eg. healthcare workers and household members of symptomatic patients who are potentially COVID positive). No symptoms of COVID infection at the time of enrollment. Potential or definite exposure to SARS-CoV-2 virus without symptoms of upper respiratory infection (smell loss, taste loss, fever, myalgia, cough, nasal congestion, runny nose, shortness of breath). All consent and testing will occur on a phone/tablet app in the participant's home.
  Interventions: Device: AROMHA Longitudinal Smell Test
- Participants with a confirmed COVID-19 infection or related smell loss: Individuals who tested positive for SARS-CoV2 by an objective PCR or antigen test will be recruited to evaluate smell function weekly over 3 months. All consent and testing will occur on a phone/tablet app in the participant's home.
  Interventions: Device: AROMHA Longitudinal Smell Test
- PASC: Known history of CSD (chemosensory dysfunction) associated with a COVID-19 infection characterized in Dr.Lora Bankova's clinical study (MGB) .
  Interventions: Device: AROMHA Longitudinal Smell Test

INTERVENTIONS:
Device: AROMHA Longitudinal Smell Test — The AROMHA Longitudinal Smell Test is a self-administered, at-home smell test intended for use as a screening test by asymptomatic individuals to help prevent exposure to and spread of SARS-CoV-2, the virus that causes COVID-19, through a serial testing approach. The device consists of six versions of a smell card, each containing three unique odors.

SUMMARY:
The purpose of this study is to learn more about how to better track smell recovery in people who have been infected with the SARS-CoV-2 virus (which causes COVID-19). Many people who have been infected by this virus develop changes in their sense of smell (olfaction). We are interested in measuring smell function objectively via smell cards that test odor intensity, identification, and discrimination. Objective and precise olfactory testing that can be performed in the convenience of one's home will help identify people with smell loss after infection by SARS-CoV-2. We will use results from this test to better understand the relationship between SARS-CoV-2 infection and recovery of olfactory function and to learn whether the AROMHA longitudinal smell test is a reliable olfactory function tracking tool to quantify smell loss in the context of COVID infection. These results may inform the design of therapeutic clinical trials to accelerate the recovery of smell function.

ELIGIBILITY:
For anosmic patients/healthy controls:

Inclusion criteria

1. Known anosmia (for anosmic patients only)
2. Age greater than or equal to 18
3. Access to phone, tablet or computer connected to the internet.

Exclusion criteria

1. Known odor-evoked adverse effects, e.g. asthma.

For asymptomatic participants:

Inclusion criteria

1. No symptoms of COVID infection at the time of enrollment.
2. Age greater than or equal to 18
3. Access to phone, tablet or computer connected to the internet.

Exclusion criteria

1. Known odor-evoked adverse effects, e.g. asthma.

For participants with COVID-19-related smell loss:

Inclusion criteria

1. Past infection of SARS-CoV-2 virus as validated by a previous PCR or antigen test
2. Age greater than or equal to 18
3. Access to phone, tablet or computer connected to the internet.

Exclusion criteria

1. Known odor-evoked adverse effects, e.g. asthma.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Diagnosis of Anosmia
  2. Healthy controls
  3. Asymptomatic patients
  4. Participants with COVID-19-related smell loss
  5. PASC with persistent smell loss
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Aromha Longitudinal Smell Test | 12 weeks
  The Aromha Smell Test is a battery of 18 odors across 6 smell cards. The subject smells each of the 3 scents per card to determine smell intensity, identification, and discrimination. Increased number of correct responses indicates better sense of smell. We will evaluate previously diagnosed anosmic patients.
Aromha Longitudinal Smell Test | 12 weeks
  The Aromha Smell Test is a battery of 18 odors across 6 smell cards. The subject smells each of the 3 scents per card to determine smell intensity, identification, and discrimination. Increased number of correct responses indicates better sense of smell. The subject's scores on the longitudinal olfactory tests will be compared to the self-reported COVID test results (SARS-CoV-2 negative or positive) of asymptomatic and symptomatic individuals.

SECONDARY OUTCOMES:
Brief Smell Identification Test (BSIT) | 12 weeks
  The BSIT is a battery of 12 odors with a score range from 0-12. Higher scores indicate a better sense of smell. We will evaluate previously diagnosed anosmic patients and healthy asymptomatic controls.

OTHER OUTCOMES:
Comparison of Aromha Longitudinal Smell Test results with upper respiratory illness | 12 weeks
  To compare results of the Aromha Longitudinal smell test with test results of upper respiratory illnesses.
Comparison of Aromha Longitudinal Smell Test results with vaccination status | 12 weeks
  To compare results of the Aromha Longitudinal smell test with self-reported vaccination status.

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Albers, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We will be sharing the results from the smell test, the answers in the demographic questionnaire, and the PCR results in a de-identified manner.
Supporting Information: CSR
Time Frame: The data will be available indefinitely and will be updated every 3 months. Our first data set will be shared in December of 2021.
Access Criteria: This study is part of the NIH RADx program, which requires sharing of de-identified participant data with a central data coordination center (RADx Data Hub). We will be sharing this information through the NIH dbGAP protocol.